CLINICAL TRIAL: NCT05091203
Title: Vitamin D as a Prognostic Marker on Assisted Reproductive Technologies Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa Adel Hanafy, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Vitamin D and IVF
Record Dates: First submitted 2021-10-02; First posted 2021-10-25 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Role of Vitamin D in IVF for Better Outcome
Keywords: ICSI- Vitamin D- BMP-15 protein
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Sham Comparator): Control group in which vitamin D was not administrated.
  Interventions: Drug: Vitamin D
- Study group (Active Comparator): Study group in which Vitamin D was administered
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — To investigate role of vitamin D in follicular maturation and number of mature follicles which help in the success of IVF procedure

SUMMARY:
Studying the effect of Vitamin D administration on assisted reproductive outcomes in women undergoing Intra Cytoplasmic Sperm Injection (ICSI) by giving a dose of vitamin D and determining the effect of this dose on both the quality embryos, implantation and ongoing pregnancy rate.

DETAILED DESCRIPTION:
1. Ninty women will include in the study. All patients will be treated with gonadotropin releasing hormone (GnRH) agonist "Decapeptyl" 0.1 mg subcutenoussubcutaneous "FeringFerring, Germany" and vitamin D (D- Dep) from day 20 of the preceding cycle till the day of HCG administration for preparation of ICSI.
2. Controlled ovarian hyper stimulation will be done with Gonal F "recombinant FSH", starting from day 3 of the stimulation cycle according to the standard protocol of the center. The dose is calculated according to the ovarian reserve, age as the BMI.
3. HCG and Vitamin D will be given when one or more of the growing follicles reaching 17 mm of diameter or more.
4. Ovum pickup was done guided by the transvaginal ultrasonography 34-36 hours after HCG administration. Follicular fluid and blood sample were obtained at the time of ovum pickup for ICSI/IVF.
5. This prospective randomized case control trial will include 90 women who will be allocated IVF/ICSI. They will be sub divided into a study and a control group; each group will include 45 women.

ELIGIBILITY:
Inclusion Criteria:

1. Age is between 20-40 years old.
2. Non PCOS patient.
3. With no previous or current evidence of OHSS (number of oocyte between 5-15 oocytes)
4. Normal Prolactin level.
5. No other endocrinological abnormality including thyroid disorder or diabetes.
6. Within normal ovarian reserve AMH(1-3) ng/ml No evidence of endometriosis.
7. No other medical or surgical diseases.

10-Careful history, general and local examination, abdominal and vaginal ultrasonography and basal haematological and chemical investigations were done

to exclude any other abnormalities which can interfere with the result of the current study.

Exclusion Criteria:

1. Women older than 35 years of age or younger than 20 years old
2. Women with polycystic ovary syndrome PCOS (as defined according to the Rotterdam criteria)
3. Women who were diagnosed to have endometriosis within the last 1 year.
4. Women with ovarian hyper stimulation syndrome (OHSS).
5. Sever male factor infertility with immotile sperm which may affect embryo development
6. poor responder patient .

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Determine the level of Vitamin D in serum and follicular fluid in ng/ml | Stimulated Cycle a bout one month
  Determine the level of Vitamin D in serum and follicular fluid in stimulated cycle for IVF/ICSI in normal responder women and comparison its level between study group (in which Vitamin D was administered) and control group ( in which vitamin D was not administrated) and its effect on oocyte quality by the use of ELISA test
Determine the level of BMP-15 in follicular fluid | Stimulated Cycle within one month
  2- Determine the level of BMP-15 in follicular fluid in stimulated cycle for IVF/ICSI in normal responder women and comparison its level between study group(in which Vitamin D was administered) and control group ( in which vitamin D was not administrated) and its effect on oocyte quality by Western Plot test

SECONDARY OUTCOMES:
To find if there is a correlation between serum and follicular fluid level of Vitamin D in the same patient. | Stimulated Cycle within one month
  After supplementation of vitamin D we will specify if there is a relation between serum and follicular fluid level of vitamin D in the same patient
4- To find if there is a relation between vitamin D and BMP 15 levels and other hormones like AMH, FSH, E2, TSH and prolactin | Stimulated Cycle within one month
  Determin the relation between vitamin D supplementation and other hormones

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt